CLINICAL TRIAL: NCT05474833
Title: Effect of Embryo Viability and Re-expansion After Thawing in Blastocyst Stage Embryos on Pregnancy Outcomes: Prospective Cohort Study
Brief Title: Assesment of Embryo Viability and Re-expansion After Thawing in Blastocyst Stage Embryos
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, ŞAFAK OLGAN, associate professor, Akdeniz University
Other Study IDs: 49849694
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Infertility
Keywords: Embryo morphology; Embryo re-expansion; Frozen- thawed embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective study, the possible effects of embryo viability and degree of blastocele re-expansion on pregnancy outcomes before vitrified/thawed blastocyst transfer will be evaluated.

DETAILED DESCRIPTION:
Thanks to the advances in embryo vitrification technologies in recent years, high embryo viability can be achieved after thawing, and live birth rates increase after the transfer of these embryos.

Embryo morphology is an essential criterion used to predict embryo viability. Blastocysts endure several morphological challenges during vitrification and thawing, including blastocele collapse, cell collapse, and subsequent rehydration. Blastocysts usually collapse immediately after thawing. Because of these morphological changes, cell damage and loss may occur, and morphological integrity may be impaired.

Considering that implantation results may be affected due to supraphysiological high estrogen and progesterone levels due to multi follicular development in the ovaries during fresh embryo transfers, the study is planned to be conducted only in patients who have undergone artificial endometrial preparation with hormone replacement therapy. Only embryos frozen at the blastocyst stage (day 5) will be included in the study.

After embryo thawing, an experienced embryologist will evaluate embryo viability and expansion and record it in the system. Approximately 2 hours after the indicated procedure (just before embryo transfer), embryo viability and degree of re-expansion will be re-evaluated by the 2nd experienced Embryologist. The evaluation results of both embryologists (embryo viability and re-expansion streams) will be known only to the primary clinician (Assoc. Prof. Şafak Olgan). Pregnancy results will be learned nine days after embryo transfer, In ultrasonography evaluation three weeks after a positive pregnancy result, a clinical pregnancy will be considered in patients with fetal heartbeat, and morphological differences between the pregnant and non-pregnant groups will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years
* Frozen- thawed embryo transfer cycles
* Only the cycles prepared artificially with hormone replacement therapy.
* Embryos with Day 5 (1CC and higher quality)

Exclusion Criteria:

* Embryos at the cleavage stage (D3)
* Patients for whom embryo viability and expansion were not evaluated single-blindly by two different embryologists

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients underwent infertility treatment
Study Population: Women between the ages of 18 and 40 who underwent IVF treatment
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Three weeks after each positive pregnancy test result
  In ultrasonography evaluation three weeks after a positive pregnancy result, a clinical pregnancy will be considered in patients with a fetal heartbeat.

SECONDARY OUTCOMES:
Positive β-hCG results | Nine days after each embryo transfer
  Positive β-hCG results nine days after embryo transfer.
The effect of re-expansion degrees and viability of embryos on pregnancy | Three weeks after each positive pregnancy test result
  The correlation between positive pregnancy results and the degree of embryo re-expansion/collapse in transfer after embryo thawing will be determined.
Optimal time between two assessments of expansion | About 2 hours between thawing and transfer
  The optimal expansion assessment time between thaw and embryo transfer will be determined. The evaluation time interval with the best pregnancy rates will be defined as optimal.

CONTACTS AND LOCATIONS:
Overall Officials: ŞAFAK OLGAN, 1, Principal Investigator — Akdeniz University; ARİF C ÖZSİPAHİ, 2, Study Chair — Akdeniz University; SEFA M CEYLAN, 2, Study Chair — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)